CLINICAL TRIAL: NCT02361177
Title: Role of Oxytocin in Telling and Detecting Lies
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug not available
Sponsor: University of Texas at Austin (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2013-11-0033
Record Dates: First submitted 2015-02-05; First posted 2015-02-11 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Dyssocial Behavior
MeSH Terms: conditions — Antisocial Personality Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxytocin (Experimental): Intranasal 24 IU oxytocin self-administration.
  Interventions: Drug: Oxytocin
- placebo (Placebo Comparator): Intranasal placebo. 125 mg of 0.5% cholorobutanol to 50 ml saline, with approximately 5 pH. The solution will then be sterilized using a 0.22 micron filter.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Intranasal oxytocin is hypothesized to amplify the influence of social norms on unethical behavior.
  Other Names: syntocinon

SUMMARY:
The investigators are interested in the impact of intranasal oxytocin in unethical behavior.

DETAILED DESCRIPTION:
The objective of this project is to further explore the role of oxytocin in moral judgment and ethical behavior. Oxytocin is a peptide hormone produced in a variety of hypothalamic neurons. It is released into the brain or brought into general circulation through sensory stimuli in a pulsatile fashion. In social psychology research, oxytocin is hypothesized to coordinate both the causes and effects of positive social interactions in a biofeedback loop.

ELIGIBILITY:
Inclusion Criteria:

* Male

Exclusion Criteria:

* _____ _____BP > 130/85, HRT > 95 (can be included at discretion of study physician/designee)

  * _____History of seizures
  * _____Neurological Disorder
  * _____Current psychiatric disorder
  * _____Previous psychiatric disorder (can be included at discretion of PI)
  * Date last episode (if > 1 year, include; if <1 year, at discretion of PI)
  * _____Current use of psychoactive drugs
  * _____Previous use of psychoactive drugs (can be included at discretion of PI) _____Date last medicated_____ _____Type of medication___________________________________
  * _____Current use of anticoagulants
  * _____Current use of corticosteroids
  * _____Previous head trauma (can be included at discretion of PI)
  * _____Alcoholism or substance abuse
  * _____Carcinoma of the breast or prostate
  * _____Renal or Hepatic diseases
  * _____Chronic lung diseases
  * _____Cancer
  * _____Liver problems
  * _____Hypertension/Cardiac diseases
  * _____Cardiovascular Disease
  * _____Nephritis
  * _____Diabetes (use of insulin) /Obesity
  * _____Endocrine disease or malignancy
  * _____Asthma (can be included as discretion of study physician/designee, if episodes are infrequent, nonmedicated, and no active problems at time of study)
  * Medication
  * Frequency of episodes____ _____Date of last episode_____
  * _____Migraines(can be included as discretion of study physician/designee, if episodes are infrequent, nonmedicated, and no active problems at time of study)
  * Medication _____Frequency of migraines_____ _____Date of last migraine_____
  * _____High levels of physical contact with women or children

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Unethical behavior | 130 minutes
  To measure unethical behavior, we will calculate whether participants took more money than they actually earned on a problem-solving task.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Josephs, PhD, Principal Investigator — utaustin

REFERENCES:
- [Result] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222